CLINICAL TRIAL: NCT04113772
Title: Orfadin and Nitinosine Study
Brief Title: Bio Equivalency 20 Mgm Orfadin and 20 Mgm of Nitisonine
Acronym: Orfadin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sutphin Drugs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Global CRO Orfadin
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Hereditary Tyrosinemia, Type I
MeSH Terms: conditions — Tyrosinemias | interventions — nitisinone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orfandin .5 mgm/kg mgm bid (Active Comparator): Two participant will receive .5 mgm/kg mgm of orfadin
  Interventions: Drug: Orfadin
- Nitinosine .5 mgm/kg bid (Experimental): Two participant will receive .5 mgm/kg of nitinosine
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — Measure bio equivalency/efficacy of nitinosine and orfadin
  Arms: Nitinosine .5 mgm/kg bid
Drug: Orfadin — Orfadin
  Arms: Orfandin .5 mgm/kg mgm bid

SUMMARY:
he purpose of this study is to determine whether Nitisinone 10 mg Tablets (Test Product are bioequivalent to the reference product Orfadin 10 mg

DETAILED DESCRIPTION:
Detailed Description:

The specific aim is to conduct a randomized, single dose, three-period crossover bioequivalence study in at least 18 healthy male and female subjects at a single study center to evaluate the in vivo performance of two formulations of Nitisinone 10 mg and the reference product Orfadin under fasting.

A total of 4 healthy female and male volunteers (age 18 to 55 years old) will be entered into the study. Volunteers will be determined to be free of significant medical conditions as assessed by medical history, physical examination, and blood and urine tests. Volunteers will be randomly allocated to a treatment sequence, before administration of investigational nitinosine

Determination of succinylacetone (SA) in blood (serum/plasma) and/or urine will be performed. Results from samples analyzed at the central laboratory, including determination of nitisinone, will be used in the evaluation of pharmacokinetics, efficacy and safety during the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* All HT-1 patients receiving Orfadin treatment are eligible for entry.
* Male and female patients of all ages diagnosed with HT-1.
* Stable lab values, including liver values <2 ULN (ALP, ALT, AST, bilirubin, INR).
* Women of childbearing potential willing to use adequate contraception
* Signed informed consent/assent.

Exclusion Criteria:

* Any medical condition which in the opinion of the investigator makes the patient unsuitable for inclusion.
* Enrollment in another concurrent clinical interventional study within three months prior to inclusion in this study.
* Pregnant women.
* Lactating women. .Known hepatitis B, hepatitis C or HIV infection.
* Foreseeable inability to cooperate with given instructions or study procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Succinylacetone level | 8 weeks
  Succinylacetone level will be measured every 2 weeks for eight weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Lifein Multi-Specialty Hospital, Navsari, Gujarat, India

IPD SHARING:
Plan to Share IPD: No